CLINICAL TRIAL: NCT06178653
Title: Examining the Effects of Trunk Control Training and Pulmonary Rehabilitation Program in Children With Spinal Muscular Atrophy
Brief Title: Two Different Treatment Modalities in Patients With Spinal Muscular Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, gorkem ata, Physiotherapist MSc./Lecturer, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-198
Record Dates: First submitted 2023-12-09; First posted 2023-12-21 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2023-01

CONDITIONS: Muscular Atrophy, Spinal
Keywords: Spinal muscular atrophy; Pulmonary rehabilitation; Trunk control; inspiratory muscle training
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulmonary Rehabilitation Group (Experimental): The program will be carried out 5 days a week, 2 times a day for 8 weeks, one day in the clinic under the supervision of the researcher, and the other four sessions in the home under the supervision of the caregiver. Caregivers will also be taught respiratory rehabilitation techniques to apply at home.
  Pulmonary Rehabilitation Training Program consists of diaphragmatic breathing, Pursed-lip breathing, and segmental breathing.
  Inspiratory muscle training: In our research, IMT will be performed in a sitting position using a handheld threshold valve device (Orygen Inspiratory Valve) that offers an adjustable inspiratory resistance via a spring-loaded valve with variable pressure load adjustment from 0-70 cmH2O. Inspiratory muscle training will be applied by calculating 30% of the maximal inspiratory pressure (MIP). During weekly clinic visits, the MIP value will be recalculated and the current threshold pressure value will be determined.
  Interventions: Other: Pulmonary Rehabilitation
- Trunk Control Training Group (Experimental): The program will be carried out 3 days a week, with pulmonary rehabilitation in each session, for a total of 45-60 minutes, for 8 weeks. The training of children whose evaluations are completed will begin after individually structured pulmonary rehabilitation and trunk control training programs are created. The content of pulmonary rehabilitation will consist of diaphragmatic breathing, pursed-lip breathing, segmental breathing, and IMT. Exercises and activities for trunk muscle activation, pelvic control, and proximal stabilization will be used together with trunk and gluteal muscle strengthening exercises. The intensity and level of exercises will be increased gradually. Body control work will first start on hard ground and then continue on soft ground and dynamic surfaces. All trunk control training will be applied actively or actively assisted.
  Interventions: Other: Pulmonary Rehabilitation; Other: Trunk Control Training

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Pulmonary rehabilitation consists of diaphragmatic, pursed-lip, and segmental breathing techniques, and also included inspiratory muscle training (will adjust 30% of maximal inspiratory pressure value)
Other: Trunk Control Training — Trunk Control Exercises will be based on the neurodevelopmental process. Exercises will progressively include activities such as stretching, turning, etc. while sitting on different surfaces (firm/soft).
  Arms: Trunk Control Training Group

SUMMARY:
Spinal Muscular Atrophy (SMA) is a severe neuromuscular disorder characterized by the degeneration of alpha motor neurons in the spinal cord, resulting in progressive muscle atrophy and weakness, particularly in proximal and axial muscles. SMA causes respiratory muscle weakness, recurrent infections, and nocturnal hypoventilation, contributing significantly to morbidity and mortality. Children with SMA often display respiratory and trunk muscle weakness compared to healthy controls. Our project aims to investigate the impact of pulmonary rehabilitation, including inspiratory muscle training, along with trunk control exercises in children with SMA. The study will include 40 SMA patients aged 5-18, with maximum inspiratory capacity below 60 centimeters of water (cmH2O), and the ability to sit unsupported for more than 5 seconds. The participants will be randomly assigned to two groups: Pulmonary Rehabilitation Group (Group 1, n=20) and Trunk Control Training Group (Group 2, n=20). Group 1 will undergo breathing exercises and inspiratory muscle training (IMT), involving diaphragmatic, pursed-lip, and segmental breathing. IMT will be administered with a portable device, starting at appropriate resistance and consisting of 10 cycles, 10 minutes each, once a day, with designated rest intervals. Also applied by calculating 30% of the maximal inspiratory pressure (MIP). During weekly clinic visits, the MIP value will be recalculated and the current threshold pressure value will be determined. In Group 2, alongside pulmonary rehabilitation, children will engage in trunk control exercises, progressively increasing in difficulty, focusing on pelvic control, proximal stabilization, and strengthening trunk and gluteal muscles. All interventions will be performed in front of a mirror. At the end of the 8-week intervention, MIP and Maximal Expiratory Pressure (MEP) will be used to measure respiratory muscle performance, spirometry will be used to monitor lung volume changes, and Peak Cough Flow will be used to evaluate the effectiveness of cough. The Trunk Control Measurement Scale, the Revised Upper Extremity Module, and the Children's Quality of Life Scale will assess trunk control, upper extremity functions, and quality of life, respectively. The Hammersmith Functional Motor Scale will assess gross motor functions and the Zarit Caregiver Burden Scale will inquire about familial factors affecting the child.

DETAILED DESCRIPTION:
Spinal Muscular Atrophy (SMA) is a severe neuromuscular disease characterized by degenerating alpha motor neurons in the spinal cord, resulting in progressive and predominantly proximal and axial muscle atrophy and weakness. Its incidence is 1 in 6000 or 10000 live births. The severity of the disease is highly variable. It causes respiratory muscle weakness, recurrent respiratory tract infections, and impaired cough with nocturnal hypoventilation in children with SMA, and is one of the leading causes of morbidity and mortality. In addition to respiratory muscle weakness, children with SMA exhibit less trunk and neck muscle activity compared to healthy controls. The aim of our project is to examine the effects of pulmonary rehabilitation practices and trunk control training combined with pulmonary rehabilitation on respiratory parameters in children with SMA. Forty SMA patients aged 5-18 years, with a maximal inspiratory capacity of less than 60 centimeters of water (cmH2O), and who can sit without support for more than 5 seconds will be included in the project. Children with SMA will be randomly divided into 2 groups. Group 1 will be the Pulmonary Rehabilitation Group (n=20), and Group 2 will be the Trunk Control Training Group (n=20). Children in group 1 will receive breathing exercises and inspiratory muscle training interventions. Breathing exercises will consist of diaphragmatic breathing to increase the efficiency of inspiration and pursed lip breathing to improve oxygenation by increasing ventilation. In addition, during segmental breathing, pressure applied by hand or with the help of a belt will provide proprioception and better expansion of the relevant regions. Inspiratory muscle training will be performed with the help of a portable device. The inspiratory muscle training program will begin at appropriate resistance and consist of a total of 10 cycles once a day, 10 minutes each with one-minute pauses in between, with 20-second pauses in between. During the pulmonary exercises, the oxygen levels of the children will be monitored with a pulse oximeter device attached to the participants' toes. In addition to pulmonary rehabilitation, the children in group 2 will perform trunk control exercises of increasing difficulty, which use a combination of exercises and activities for pelvic control and proximal stabilization, and trunk and gluteal muscle strengthening exercises. All interventions will be performed in front of the mirror. Children's fatigue levels will be determined according to the perceived exertion level. The intervention of both groups will last 8 weeks. Evaluation parameters will be applied before interventions begin and at the end of 8 weeks. Respiratory performance and respiratory muscle strength, which are among the primary measurement parameters, are measured by Maximal Inspiratory Pressure and Maximal Expiratory Pressure; lung capacities will be evaluated by using a spirometer device where pulmonary function tests are applied, and the effectiveness of cough will be evaluated by measuring the Peak Cough Flow value. Trunk Control Measurement Scale in the evaluation of trunk control; Revised Upper Extremity Module for evaluation of upper extremity functions. In the examination of changes in lung volumes, a data record will be created using chest radiography. Hammersmith Functional Motor Scale in the evaluation of gross motor functions; The Children's Quality of Life Scale will be used to evaluate the quality of life of the cases; familial factors affecting children will be questioned with the Zarit Caregiver Burden Scale.

ELIGIBILITY:
Inclusion Criteria:

* Those with genetic documentation of 5q spinal muscular atrophy (SMA) homozygous gene deletion, mutation, or compound heterozygote and who have been clinically diagnosed with SMA,
* Those between the ages of 5-18,
* Maximum inspiratory capacity is less than 60 cmH2O,
* Children who can sit unsupported for at least 5 seconds and who have no or 3 weeks of acute reversible events affecting the upper respiratory tract.

Exclusion Criteria:

* Having had upper extremity and spine surgery,
* Having other orthopedic and neurological problems,
* Having cognitive impairments that may prevent understanding simple verbal commands,
* Having visual or auditory disabilities,
* Premature birth

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Inspiratory Muscle Strength | 8 weeks
  Inspiratory Muscle Strength will be assessed by the Maximal Inspiratory Pressure (MIP). For MIP measurement, participants will be asked to perform maximum inspiration starting from the residual lung volume following maximum expiration to the total lung capacity.
Expiratory Muscle Strength | 8 weeks
  Expiratory Muscle Strength will be assessed by the Maximal Expiratory Pressure (MEP). For MEP measurement, participants will be asked to exert maximum expiratory effort from total lung capacity to residual volume. Pressure thresholds sustained for at least 1 second will be recorded. The highest pressure value of these maneuvers, expressed in cmH2O, will be recorded.
Pulmonary Function Test | 8 weeks
  Participants will be in a sitting position during spirometric measurement in accordance with the standards and recommendations of the American Thoracic Society and European Respiratory Society statement. Forced vital capacity (FVC), volume of air exhaled in the 1st second of forced expiration (FEV1), FEV1/FVC ratio, peak expiratory flow (PEF) values of the participants will be measured through spirometric (Spirobank MIR, Italy) measurement. At least three successful spirometric assessments will be recorded. FVC is the volume of air exhaled rapidly and forcefully following deep inspiration. PEF value is measured by maximum inspiration followed by maximum expiration. It usually correlates with FEV1 measurements. In the interpretation of spirometric tests, information can be obtained about the type and severity of respiratory dysfunction by looking at the shape and numerical parameters of the flow-volume and time curve.
Effectiveness of Cough | 8 weeks
  The effectiveness of the cough will be evaluated with a Peak Flow meter. This value provides us with information about the expiratory muscles. To evaluate the ability to cough without assistance, the patient is asked to cough as hard as possible into a small handheld device called a peak flow meter (ExpiritePeak Flow Meter DL-F03) while in a sitting position. This measured value is called peak cough flow (PCF). These values will provide an indication of the patient's disease progression, ability to clear secretions, and risk of developing respiratory complications. PCF is applied to children over the age of 4-8. The expected value in healthy individuals is PCF ≥ 360 L/minute. The fact that this value is 270 L/minute in children with DMD, another neuromuscular muscle disease, shows that participants have adequate cough. A PCF value falling below 160 L/minute indicates inadequate airway clearance. Absolute values will be determined by selecting the largest of three consecutive trials.

SECONDARY OUTCOMES:
Trunk Control | 8 weeks
  Trunk Control will be assessed by Trunk Control Measurement Scale. Children's trunk control levels will first be determined according to the Trunk Control Measurement Scale (TCMS), which was developed for children with cerebral palsy. The TCMS consists of 15 items that evaluate 2 different parameters related to trunk control; One of the parameters is static sitting balance and the other is dynamic sitting balance. It evaluates not only trunk control but also trunk compensation during limb movements. Within dynamic sitting balance, balance parameters in reaching and reaching are also evaluated. Total scores range from 0 to 58, with higher scores indicating good trunk control.
Upper Extremity Functions | 8 weeks
  Upper Extremity Functions will be assessed by Revised Upper Limb Module for Spinal Muscular Atrophy. The revised upper extremity module for SMA contains 19 items and is evaluated out of a total of 37 points. The first item is not included in the scoring, and the remaining 18 items are evaluated between 0-2 points, except for item I, and only item I is evaluated between 0-1 points. The module is calculated on a total of 37 points, higher scores indicate better upper extremity function.
Gross Motor Function | 8 weeks
  Gross Motor Function levels will ve assessed by the Hammersmith Functional Motor Scale. It measures the motor function changes of children with SMA who can and cannot walk. It consists of 33 items that indicate the capacity to perform motor functions such as sitting on a chair without support, lying face down or rolling over, lifting the head from the prone position, and crawling. Each activity, categorized into items, is scored on a 3-point system with 2 points for "performs without modification", 1 point for "performs with modification/adaptation/compensation" and 0 points for "cannot perform the task". The maximum score on the scale is 66, and a higher score means better motor functions.
Quality of Life of the Children | 8 weeks
  In evaluating the quality of life of patients with SMA; Pediatric Quality of Life Questionary-Generic Core (PedsQL-GC) will be used. It questions the areas of physical health, emotional functionality, and social functionality, which are the characteristics of the state of health defined by the World Health Organization. Items are scored between 0-100. If the answer to the question is marked as never, it receives 0=100, if it is marked as rarely, it receives 1=75, if it is marked as sometimes, it receives 2=50, if it is marked as often, it receives 3=25, and if it is marked as almost always, it receives 4=0 points. The total score is obtained by adding the points and dividing by the number of items completed. If more than 50% of the scale is not filled out, the scale is not evaluated. The higher the total score, the better the health-related quality of life is perceived.
Burden of Caregiver | 8 weeks
  Caregiver burden score will be evaluated by the Zarit Caregiver Burden Interview. It was developed by Zarit, Reever and Bach-Peterson in 1980. It is a scale used to evaluate the distress experienced by caregivers of individuals in need of care. The scale, which can be completed by asking the caregivers themselves or the researcher, consists of 19 statements that determine the impact of caregiving on the individual's life. The scale has a Likert-type rating ranging from 1 to 5, such as never, rarely, sometimes, often or almost always. A high scale score indicates that the distress experienced is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol Mega University Hospital, Istanbul, Bağcılar, Turkey (Türkiye)